CLINICAL TRIAL: NCT05569109
Title: av Fistula Patency Loss as a Cause of Fistula Failure and Its Relation to Hyperphosphatemia in Chronic Hemodialysis Patients
Brief Title: av Fistula Patency Loss as a Cause of Fistula Failure and Hyperphosphatemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kerollos Refaat Labeeb, M.B.B.CH , M.Sc, Assiut University
Other Study IDs: av fistula and phosphate
Record Dates: First submitted 2022-09-27; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: AV Fistula
Keywords: hyperphosphatemia
MeSH Terms: conditions — Arteriovenous Fistula; Hyperphosphatemia | interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- av fistula patency loss with hperphosphatemia: hemodialysis patients with av fistula patency loss by doppler ultrasound and hyperphosphatemia
  Interventions: Device: doppler ultrasound
- av fistula patency loss with normal phosphate level: hemodialysis patients with av fistula patency loss by doppler ultrasound and normal phosphate level
  Interventions: Device: doppler ultrasound

INTERVENTIONS:
Device: doppler ultrasound — doppler ultrasound on arteriovenous fistula in hemodialysis patients

SUMMARY:
Assessment of arteriovenous fistula patency loss which leads to av fistula failure and its relation to high serum phosphate level in chronic hemodialysis patients.

DETAILED DESCRIPTION:
End-stage renal disease is a chronic disease requiring treatment with dialysis or renal transplantation. Patients require an adequate vascular access for hemodialysis (HD). Autologous arteriovenous fistula (AVF) is gold standard to maintain vascular access for HD . Vascular access-related complications can lead to patient morbidity and reduction of patient quality of life.The complication rate related to permanent HD vascular access remains relatively high and access related problems are responsible for 50% of the hospitalization of dialysis patients. Secondary failures are not rare and in need of adequate attention and care. Once the AVF has been placed. It is recommended that serial monitoring of the AVF should be done for long term effective function. Delays in preventing complications may lead to AVF dysfunction. However, little is known about the factors determining long term prognosis of an AVF.

Primary patency (intervention-free access survival) was defined as the interval from time of access placement to any intervention designed to maintain or reestablish patency or to access thrombosis or the time of measurement of patency. Assisted primary patency (thrombosis-free access survival) was defined as the interval from time of access placement to access thrombosis or time of measurement of patency, including intervening manipulations (surgical or endovascular interventions) designed to maintain the functionality of a patent access. Secondary patency (access survival until abandonment) was defined as the interval from time of access placement to access abandonment or time of measurement of patency, including intervening manipulations (surgical or endovascular interventions) designed to reestablish the functionality of thrombosed access .

In patients having chronic renal failure (CRF), several changes occur in bone metabolism due to the development of secondary hyperparathyroidism. There are increased calcium and phosphate release from bones to the blood, causing the deposition of calcium and phosphate in the intima-media layer of arterial wall and eventuating vascular calcification in these patients. The deposition of these electrolytes increases the risk of cerebrovascular and coronary complications as well. Thus, a decrease in the quality of fistula occurs in these tracts utilized frequently at the arteriovenous fistula (AVF) operations.

ELIGIBILITY:
Inclusion Criteria:

* adult patients more than 18 years old with end stage renal disease on regular hemodialysis using arteriovenous fistula

Exclusion Criteria:

* : patients less than 18 years, patients with peripheral artery diseases, access failure occurred within the first 2 months after fistula surgery, AVF failure was related to an infectious complication and patients with arteriovenous grafts.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - adult patients more than 18 years old with end stage renal disease on regular hemodialysis using arteriovenous fistula
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
measurement of early av fistula patency loss | baseline
  early measurement of av fistula patency loss using doppler ultrasound to decrease the fistula failure rate

SECONDARY OUTCOMES:
measurement if there is a relation between fistula patency loss and hyperphosphatemia | baseline
  analysis if a high serum phosphate level leads to arteriovenous fistula patency loss

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Assiut U, Asyut, Egypt

REFERENCES:
- [Background] Tuysuz ME, Dedemoglu M. Calcium phosphate product level as a predictor for arteriovenous fistula re-operations in patients with chronic renal failure. Vascular. 2019 Jun;27(3):284-290. doi: 10.1177/1708538118814611. Epub 2018 Nov 21. PMID 30463499
- [Background] Cozzolino M, Gallieni M, Brancaccio D. The mechanisms of hyperphosphatemia-induced vascular calcification. Int J Artif Organs. 2008 Dec;31(12):1002-3. doi: 10.1177/039139880803101203. PMID 19115191
- [Background] Manne V, Vaddi SP, Reddy VB, Dayapule S. Factors influencing patency of Brescia-Cimino arteriovenous fistulas in hemodialysis patients. Saudi J Kidney Dis Transpl. 2017 Mar-Apr;28(2):313-317. doi: 10.4103/1319-2442.202759. PMID 28352013
- [Background] MacRae JM, Dipchand C, Oliver M, Moist L, Lok C, Clark E, Hiremath S, Kappel J, Kiaii M, Luscombe R, Miller LM; Canadian Society of Nephrology Vascular Access Work Group. Arteriovenous Access Failure, Stenosis, and Thrombosis. Can J Kidney Health Dis. 2016 Sep 27;3:2054358116669126. doi: 10.1177/2054358116669126. eCollection 2016. PMID 28270918
- [Background] Moghazy KM. Value of color Doppler sonography in the assessment of hemodialysis access dysfunction. Saudi J Kidney Dis Transpl. 2009 Jan;20(1):35-43. PMID 19112217
- [Background] Huijbregts HJ, Bots ML, Wittens CH, Schrama YC, Moll FL, Blankestijn PJ; CIMINO study group. Hemodialysis arteriovenous fistula patency revisited: results of a prospective, multicenter initiative. Clin J Am Soc Nephrol. 2008 May;3(3):714-9. doi: 10.2215/CJN.02950707. Epub 2008 Feb 6. PMID 18256379